CLINICAL TRIAL: NCT01583166
Title: Voiding Function After Mid-Urethral Slings With and Without Local Anesthetic: Randomized Controlled Trial
Acronym: URINE&ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Michael Flynn, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: 14197
Record Dates: First submitted 2012-04-19; First posted 2012-04-23 (Estimated); Results first posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-10

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Bupivacaine; Sodium Chloride; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine + epinephrine (Active Comparator)
  Interventions: Drug: Bupivacaine; Drug: Epinephrine
- Saline + epinephrine (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bupivacaine — 10ml 0.5% bupivacaine
  Other Names: Marcaine
  Arms: Bupivacaine + epinephrine
Drug: Saline — 10ml 0.9% sodium chloride
  Other Names: Sodium Chloride
  Arms: Saline + epinephrine
Drug: Epinephrine — 1:200,000 epinephrine
  Arms: Bupivacaine + epinephrine

SUMMARY:
The purpose of this study is to determine if there is a difference in post-operative voiding function between subjects receiving local anesthetic and those receiving placebo at the time of mid-urethral sling placement. The secondary objective is to evaluate pain after the procedure in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo mid-urethral sling for incontinence without concomitant procedures

Exclusion Criteria:

* Undergoing procedure in addition to the sling
* Not competent to give consent
* Using intermittent self catheterization pre-operatively
* Known allergy to local anesthetic
* Undergoing spinal anesthesia for the procedure
* Prisoners
* Non-English speaker
* Under 18 years of age
* Has a condition that would contra-indicate the use of local anesthetic or epinephrine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Flynn, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Duenas-Garcia OF, Patterson D, De la Luz Nieto M, Leung K, Flynn MK. Voiding Function After Midurethral Slings With and Without Local Anesthetic: Randomized Controlled Trial. Female Pelvic Med Reconstr Surg. 2017 Jan/Feb;23(1):56-60. doi: 10.1097/SPV.0000000000000343. PMID 27682748

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with stress incontinence or stress-predominant mixed urinary incontinence who were scheduled to undergo a retropubic midurethral sling with no concomitant procedures at UMass Memorial Healthcare, Inc.
  Enrollment occurred from March 2012 to June 2015 with study presented and consent sought at time of preoperative appointment.
Pre-assignment Details: 10 participants did not receive allocated intervention--patient-initiated cancellation of surgery. (Saline + Epinephrine n=6, Bupivavane + Epinephrine n=4). Midway through study, indigo carmine became unavailable and surgical team opted for phenazopyridine. Failed to obtain 6-7 hour pain score in 24 out of 80 subjects.
Groups:
- Marcaine + Epinephrine: Bupivicaine + epinephrine: 10ml 0.5% bupivicaine plus 1:200,000 epinephrine
- Saline + Epinephrine: Sodium chloride + epinephrine: 10ml 0.9% sodium chloride plus 1:200,000 epinephrine
Period: Overall Study
Arm/Group | Marcaine + Epinephrine | Saline + Epinephrine
Started | 45 | 45
Completed | 41 | 39
Not Completed | 4 | 6
Not completed — Withdrawal by Subject | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Marcaine + Epinephrine | Saline + Epinephrine | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: all subjects were included in the baseline assessments
  the final numbers in the results section differ due to subject withdrawal or drop out
  years | 46.0 (11.6) | 50.5 (11.1) | 48.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 39 | 80
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: 45 randomized to each, number analyzed differs due to participant withdrawal
  Participants
    United States | 41 | 39 | 80
Visual Analog Scale for Pain: Preoperative [Mean (Standard Deviation); unit: Units on a Scale] — Participants were asked to report on pre-operative level of pain using a Visual Analog Scale, The scale is participant reported and ranged form 0 representing no pain to 10 representing unbearable pain.
  Units on a Scale | 0.0 (1) | 0.0 (1.4) | 0.0 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Passed the Voiding Trial After a Midurethral Sling
Description: Study team assessment of whether the use of local anesthetic has any affect on the percentage of patients who pass their post-operative bladder challenge. This is determined by their voided volume and post-void residual.
Time Frame: 2 weeks
Population: Passed void trial
Measure: Count of Participants; unit: Participants
Arm/Group | Marcaine + Epinephrine | Saline + Epinephrine
Number analyzed (Participants) | 41 | 39
Participants | 31 | 32

2. Secondary Outcome: Post-operative Pain Scores at 2-3 Hours Post op
Description: Visual analog score at 2 hours post op will be compared in the two groups. The scale ranges from 0 (no pain) to a maximum of 10 (unbearable pain)
Time Frame: 2-3 hours
Population: Please notice that the number of subjects is different because we only analyzed the pain scores from the subjects who were randomized and had the surgery. We also had some missing pain scores
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Marcaine + Epinephrine | Saline + Epinephrine
Number analyzed (Participants) | 41 | 39
units on a scale | 3 (2) | 2.9 (2.1)
Statistical Analysis 1: Comparison: Marcaine + Epinephrine vs Saline + Epinephrine; Test type: Other; p = 0.837, Fisher Exact

3. Secondary Outcome: Post-operative Pain Scale at 6-7 Hours Post op
Description: Visual analog score at 6 hours post op will be compared in the two groups. The scale ranges from 0 (no pain) to a maximum of 10 (unbearable pain)
Time Frame: 6-7 hours
Population: Study team failed to obtain 6-7 hour pain score for 24 out of the 80 participants. The overall number of participants analyzed reflects this occurence.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Marcaine + Epinephrine | Saline + Epinephrine
Number analyzed (Participants) | 29 | 27
units on a scale | 3.1 (1.6) | 4.1 (1.9)

4. Secondary Outcome: Visual Analog Scale for Pain: Pre-operative.
Description: Participants asked to report on pre-operative level of pain using a Visual Analog Scale. The scale is participant reported and ranges from 0 representing no pain to 10 representing unbearable pain.
Time Frame: At enrollment
Population: Please noticed that there is a discrepancy with the number of subjects. We include the data from all subjects who were randomized and had the intervention.
Measure: Mean (Standard Deviation); unit: Reported Pain Level score on VAS
Arm/Group | Marcaine + Epinephrine | Saline + Epinephrine
Number analyzed (Participants) | 41 | 39
Reported Pain Level score on VAS | 0.0 (1) | 0.0 (1.4)

ADVERSE EVENTS:
Arm/Group | Marcaine + Epinephrine | Saline + Epinephrine
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

LIMITATIONS AND CAVEATS:
Failure to obtain 6-7 hour pain score for 24/80 participants. Impact of large preponderance of slings placed by a subrapublic approach. Study not designed to examine the effect of phenazopyridine in study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No